CLINICAL TRIAL: NCT03375970
Title: Establishing the Collaborative Care Model of TCM and Western Medicine-Pediatric Atopic Dermatitis
Brief Title: Establishing the Collaborative Care Model of Traditional Chinese Medicine and Western Medicine-Pediatric Atopic Dermatitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Hung-Rong Yen, Attending physician, China Medical University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMUH106-REC2-029
Record Dates: First submitted 2017-05-26; First posted 2017-12-18 (Actual); Last update posted 2017-12-18 (Actual); Status verified 2017-04

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collaborative Care of TCM and Western Medicine (Experimental)
  Interventions: Other: TCM; Other: Western medicine
- Western Medicine (Active Comparator)
  Interventions: Other: Western medicine

INTERVENTIONS:
Other: TCM — oral chinese herb, chinese topical ointment
  Arms: Collaborative Care of TCM and Western Medicine
Other: Western medicine — oral steroid, oral antihistamine, topical steroid

SUMMARY:
In Taiwan, there are many patients suffer from pediatric atopic dermatitis. Because of the clinical characteristic of repetitive and scratchy, which will affect the patients' quality of life and lead to the medical heavy budget. TCM may play an important role in this disease and help patient to improved their health. In this project, we aim to establish a Collaborative Care Model of TCM and Western Medicine, to achieve the multiple goal in clinical treatment, research and medical training. By establishing a collaborative care model, including the Chinese medicine doctor and Western medicine doctor, nurses, pharmacists and case managers, to cooperative satisfy the patient needed in the medical service, to improve the clinical presentation, patients'quality of life, and reduce exposure to corticosteroid. Besides, we can also build a training environment and reduce medical cost in long term purpose. Furthermore, by establishing a collaborative care model, we can provide a medical education and training opportunity to educate the medical student and clinician the necessary knowledge of pediatric atopic dermatitis by caring patients and learning from clinical case. According to the above training program, we not only aim to strengthen the competitiveness of Chinese medicine doctor in Taiwan, but also make the Western medicine doctors comprehend the TCM characteristic and may find out the even more opportunity to cooperate in clinical practice. To make this collaborative care model as a beginning milestone of cooperation between Chinese medicine and Western medicine.

ELIGIBILITY:
Inclusion Criteria:

* age 0-18
* meets the Hanifin and Rajka diagnostic criteria
* SCORAD score ≧ 25

Exclusion Criteria:

* Drug abuse
* Pregnent or lactating women
* Mental or behavioral abnormalities
* Allergic to the ingredients of the test regimen
* Any potentially life-threatening disease or dysfunctional organ system l

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-05-02 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Scoring Atopic Dermatitis (SCORAD) score | week 4
  a clinical tool to assess the extent and severity of eczema

SECONDARY OUTCOMES:
36-Item Short Form Health Survey (SF-36) | week 4
  It is a 36-item, patient-reported survey of patient health.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan